CLINICAL TRIAL: NCT01003665
Title: Accuracy of the CNAP™ Monitor (Continuous Non-invasive Arterial Pressure) Versus Invasive Radial Arterial Monitoring in Surgical Patients
Brief Title: Comparison of Continuous Non-invasive Arterial Pressure (CNAP) With Invasive Arterial Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Robert Hanss, Prof. Dr. Robert Hanss, University Hospital Schleswig-Holstein
Other Study IDs: CNAP-2009-1
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intensive Care treatement: ASA status 3 or 4 patients with invasive blood pressure measurement on the intensive care unit

SUMMARY:
The purpose of this study was to compare the Continuous Non-invasive Arterial Pressure (CNAP) monitor with the gold standard of invasive arterial pressure monitoring during:

1. induction and maintenance of general anaesthesia
2. intensive care unit treatment of postoperative patients with an ASA 3 or 4 status

DETAILED DESCRIPTION:
The CNAP monitor continuously measures blood pressure using a finger cuff. It showed a good agreement to invasive blood pressure measurements during anaesthesia induction and maintenance during surgery. In critical ill patients cardiac arrhythmia is probably a confounding factor affecting accuracy and interchangeability of CNAP. As systolic arterial CNAP pressure in comparison to mean pressure shows no statistical interchangeability with invasive measurements, mean pressure should be considered when making therapy decisions.

A problem is the missing standard criterion for comparison of continuously devices with invasive pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* BMI < 35 kg.m²
* Patients capable of giving informed consent
* patients undergoing elective surgical procedures in supine position under general anesthesia
* perfusion of the examined arm evidenced by a positive Allen's test

Exclusion Criteria:

* Patients not competent or unwilling to provide informed consent
* Patients with history of neurological, neuromuscular seizure
* Patients where IBP cannula, CNAP™ finger-cuff and CNAP™ upper arm cuff cannot be placed on the same arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing major surgery or intensive care unit treatement with the need for an invasive blood pressure measurement
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Bias and percentage error of CNAP compared with invasive arterial pressure measurement | 1.) Induction of general anaesthesia. 2.) Maintanance of general anaesthesia. 3.) Intensive Care Treatement after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Markus Steinfath, Professor, Study Chair — Klinik für Anästhesiologie und Operative Intensivmedizin, UKSH Kiel; Robert Hanss, Professor, Study Director — Klinik für Anästhesiologie und Operative Intensivmedizin, UKSH Kiel
Locations (1):
- Klinik für Anästhesiologie und Operative Intensivmedizin, Universitätsklinik Schleswig-Holstein, Campus Kiel, Kiel, Germany

REFERENCES:
- [Result] Ilies C, Bauer M, Berg P, Rosenberg J, Hedderich J, Bein B, Hinz J, Hanss R. Investigation of the agreement of a continuous non-invasive arterial pressure device in comparison with invasive radial artery measurement. Br J Anaesth. 2012 Feb;108(2):202-10. doi: 10.1093/bja/aer394. Epub 2011 Dec 12. PMID 22171358
- [Derived] Ilies C, Grudev G, Hedderich J, Renner J, Steinfath M, Bein B, Haake N, Hanss R. Comparison of a continuous noninvasive arterial pressure device with invasive measurements in cardiovascular postsurgical intensive care patients: a prospective observational study. Eur J Anaesthesiol. 2015 Jan;32(1):20-8. doi: 10.1097/EJA.0000000000000136. PMID 25105850